CLINICAL TRIAL: NCT02248506
Title: Epidemiological Study About the Clinical and Microbiological Evolution of Patients Treated for an Acute Episode of Vulvovaginal Candidiasis.
Brief Title: Epidemiological Study About the Evolution of Patients Treated for an Acute Episode of Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: Gynea Laboratorios SA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GY-LAC-01-2012
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Candidiasis, Vulvovaginal
Keywords: Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis | interventions — Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clotrimazole (Other): Clotrimazole 500 mg
  Interventions: Other: Clotrimazole

INTERVENTIONS:
Other: Clotrimazole — All patients receive standard antifungal treatment for this type of infections consisting Clotrimazole 500 Single dose (standard treatment).

SUMMARY:
To determine proportion of women achieving clinical and mycological cure or have recurrences / reinfection after being treated for an acute episode of vulvovaginal candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women between 18 and 50 years
* Patients attending to the gynecologist with acute vulvovaginal candidiasis.
* Patients requiring standard treatment with clotrimazole 500 single dose and that the decision to prescribe this treatment is prior to inclusion in the study.
* Women who agree to participate in the study and has signed the informed consent sheet.

Exclusion Criteria:

* Use of any medication that may interfere significantly with study assessments.
* Pregnant or breastfeeding
* Women with signs of other genital infection
* Within 3 months after childbirth or abortion
* Patients that is expected not to attend follow-up visits

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Vaginal swab test | Baseline
  To verify diagnosis of vaginal candidiasis
Vaginal swab test | month 2
  To determine proportion of women achieving clinical and mycological cure or have recurrences / reinfection after being treated for an acute episode of vulvovaginal candidiasis
Vaginal swab test | month 3
  To determine proportion of women achieving clinical and mycological cure or have recurrences / reinfection after being treated for an acute episode of vulvovaginal candidiasis
Vaginal swab test | month 6
  To determine proportion of women achieving clinical and mycological cure or have recurrences / reinfection after being treated for an acute episode of vulvovaginal candidiasis, only those with a history of more than four episodes in a year

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Madrid, Spain